CLINICAL TRIAL: NCT02848781
Title: PAUSE-SCD: Pan-Asia United States PrEvention of Sudden Cardiac Death Catheter Ablation Trial
Brief Title: Pan-Asia United States PrEvention of Sudden Cardiac Death Catheter Ablation Trial
Acronym: PAUSE-SCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000272
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Results first posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-03

CONDITIONS: Ventricular Tachycardia (VT)
Keywords: Sudden Cardiac Death; ICD Therapy; VT Ablation
MeSH Terms: conditions — Tachycardia, Ventricular; Death, Sudden, Cardiac | interventions — Defibrillators, Implantable; Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ICD with Ablation (Experimental): Patient will receive an implantable cardioverter defibrillator (ICD) with catheter ablation and standard medical management.
  Interventions: Device: Implantable Cardioverter Defibrillator (ICD); Procedure: Catheter Ablation
- ICD Only (Active Comparator): Patient will receive an implantable cardioverter defibrillator (ICD) and standard medical management.
  Interventions: Device: Implantable Cardioverter Defibrillator (ICD)
- Ablation Only (Registry) (Active Comparator): The registry will enroll patients who refuse an implantable cardioverter defibrillator (ICD) and are thus not randomized. This arm will assess the efficacy of catheter ablation in the absence of background ICD therapy.
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator (ICD) — An ICD is a battery-powered device placed under the skin that keeps track of heart rate. Thin wires connect the ICD to the heart. If an abnormal heart rhythm is detected, the device will deliver an electric shock to restore a normal heartbeat.
  Arms: ICD Only; ICD with Ablation
Procedure: Catheter Ablation — Catheter ablation is a procedure that uses radiofrequency energy to destroy a small area of heart tissue that is causing rapid and irregular heartbeats. Destroying this tissue helps restore the heart's regular rhythm.
  Arms: Ablation Only (Registry); ICD with Ablation

SUMMARY:
The current standard of care for ventricular tachycardia (VT) includes the use of medicine called anti-arrhythmic drugs (AADs) and Implantable Cardioverter Defibrillator (ICD) therapy. These treatments are used to terminate the irregular heartbeats and bring the heart back to a normal rhythm. Catheter ablation is a procedure used to eliminate (damage) the heart cells causing the arrhythmia. Patients eligible for this may benefit from an ablation procedure in addition to an ICD to treat their VT condition or risk of developing VT. This study aims to show that treating VT with catheter ablation, if performed preemptively at the time of ICD implantation, will reduce subsequent recurrent VT, ICD shocks, and lead to improved survival.

DETAILED DESCRIPTION:
Subjects who meet inclusion/exclusion criteria will be entered into the randomized trial. Randomization will be 1:1 between control group and ablation group. Those randomized to the control group will receive ICD therapy and routine drug therapy (including antiarrhythmic drugs as indicated). Subjects randomized to the ablation group will receive ablation therapy plus ICD for ventricular tachycardia. Patients that refuse ICD therapy and undergo ablation only will be enrolled in a prospective registry.

Follow-up will be performed prior to hospital discharge for incision check and device interrogation as is standard of care. In addition, routine device and clinical follow-up will be scheduled at 1, 3, 6, 12, 18, and 24 months. Electrocardiography (ECG) will be performed pre-implant and prior to hospital discharge. Echocardiography (TTE) will be performed pre-implant and at 12 and 24 months.

Patients that refuse ICD implantation will not be randomized and will be approached for inclusion into a registry if they undergo catheter ablation without an ICD. Basic demographics and medical history will be collected from registry subjects upon enrollment. Registry subjects will receive follow-up for routine clinical care every 6 months to check on their overall status.

120 subjects will be randomized. An additional 60 subjects will enrolled into the registry.

As of the time protocol revision C changes were made (07Nov2016), 33 subjects have been randomized. There has not been any preliminary or interim analysis of any data at this point. The study-sponsor has not had any access to any clinical follow-up for the patients enrolled to date.

ELIGIBILITY:
Inclusion Criteria:

* Patient is receiving a new implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy device (CRT-D) implant that has study required programing capabilities and is appropriate for remote monitoring. Patient who has received the ICD / CRT-D within 90 days of enrollment can also be enrolled.
* Patient who has a high risk of ICD shock as shown by documented Monomorphic VT (MMVT) by one or more of the following:

  * Spontaneous MMVT
  * Inducible MMVT during electrophysiology study,
  * Inducible MMVT during noninvasive programmed stimulation study *Inducible MMVT is defined as MMVT > 30 seconds or requiring electrical termination (ATP or cardioversion)
* Patient has ejection fraction < 50% or right ventricular dysfunction
* Patient has a cardiomyopathy with structural heart disease of any cause

Exclusion Criteria:

* Any history of debilitating stroke with neurologic deficit
* ST-segment elevation myocardial infarction or previous cardiac surgery within 60 days prior to enrollment
* Patient is pregnant or nursing
* Patient has chronic New York Heart Association (NYHA) class IV heart failure
* Patient has incessant VT necessitating immediate treatment
* Patient has ventricular tachycardia/ventricular fibrillation thought to be from channelopathies
* Limited life expectancy (less than one year)
* Patient has current class IV angina
* Recent coronary artery bypass graft or percutaneous coronary intervention (< 45 days)
* Patient is currently participating in another investigational drug or device study
* Known presence of intracardiac thrombi
* Prosthetic mitral or aortic valve or mitral or aortic valvular heart disease requiring immediate surgical intervention
* Major contraindication to anticoagulation therapy or coagulation disorder
* Left Ventricular Ejection Fraction < 15%
* Patient has had a previous ablation procedure for VT, excluding remote (> 3 months) outflow tract tachycardia
* Patient has glomerular filtration rate (GFR) < 30 mL/min/1.73m2
* Patient has peripheral vascular disease that precludes left ventricular access
* Patient is thought to have idiopathic outflow VT as only VT
* Patient has a premature ventricular contraction (PVC) or VT induced cardiomyopathy that is expected to resolve with ablation and will not require an ICD
* Patient has reversible cause of VT
* Patient does not meet criteria for ICD or CRT-D

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roderick Tung, MD, Study Director — University of Chicago
Locations (12):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States
- China (6):
  - Fuwai Cardiovascular Hospital, Beijing
  - Huaxi Hospital, Chengdu
  - Guangdong General Hospital, Guangzhou
  - Sir Run Run Shaw Hospital, Hangzhou
  - Nanjing First Affiliated Hospital, Nanjing
  - PLA Shenyang General Hospital, Shenyang
- Japan (3):
  - Dokkyo Medical University, Saitama Medical Center, Saitama
  - Kyorin University Hospital, Tokyo
  - Tsukuba University, Tsukuba
- Korea University, Seoul, South Korea
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tung R, Xue Y, Chen M, Jiang C, Shatz DY, Besser SA, Hu H, Chung FP, Nakahara S, Kim YH, Satomi K, Shen L, Liang E, Liao H, Gu K, Jiang R, Jiang J, Hori Y, Choi JI, Ueda A, Komatsu Y, Kazawa S, Soejima K, Chen SA, Nogami A, Yao Y; PAUSE-SCD Investigators. First-Line Catheter Ablation of Monomorphic Ventricular Tachycardia in Cardiomyopathy Concurrent With Defibrillator Implantation: The PAUSE-SCD Randomized Trial. Circulation. 2022 Jun 21;145(25):1839-1849. doi: 10.1161/CIRCULATIONAHA.122.060039. Epub 2022 May 4. PMID 35507499
- [Derived] Kheiri B, Barbarawi M, Zayed Y, Hicks M, Osman M, Rashdan L, Kyi HH, Bachuwa G, Hassan M, Stecker EC, Nazer B, Bhatt DL. Antiarrhythmic Drugs or Catheter Ablation in the Management of Ventricular Tachyarrhythmias in Patients With Implantable Cardioverter-Defibrillators: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Circ Arrhythm Electrophysiol. 2019 Nov;12(11):e007600. doi: 10.1161/CIRCEP.119.007600. Epub 2019 Nov 8. PMID 31698933

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Not Applicable - no wash out or run-in periods.
Period: Overall Study
Arm/Group | ICD With Ablation | ICD Only | Ablation Only (Registry)
Started | 67 | 66 | 47
Completed | 60 | 61 | 47
Not Completed | 7 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ICD With Ablation | ICD Only | Ablation Only (Registry) | Total
Number analyzed (Participants) | 60 | 61 | 47 | 168
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 47 | 40 | 131
  >=65 years | 16 | 14 | 7 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 7 | 30
  Male | 44 | 54 | 40 | 138
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 60 | 61 | 47 | 168
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 2 | 1 | 0 | 3
  China | 50 | 49 | 47 | 146
  Japan | 3 | 5 | 0 | 8
  Taiwan | 5 | 6 | 0 | 11

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Recurrent VT, Cardiovascular Rehospitalization, and All-cause Mortality
Description: The primary endpoint is a composite.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | ICD With Ablation | ICD Only | Ablation Only (Registry)
Number analyzed (Participants) | 60 | 61 | 47
Participants
  Freedom from recurrent VT, cardiovascular rehospitalization, and all-cause mortality | 33 | 25 | 28
  Recurrent VT, cardiovascular rehospitalization, and all-cause mortality | 27 | 36 | 19

2. Secondary Outcome: Freedom From Recurrent VT
Description: Recurrent VT is defined as any appropriate ICD therapy (shock or ATP) or documented sustained monomorphic VT >30 seconds.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | ICD With Ablation | ICD Only | Ablation Only (Registry)
Number analyzed (Participants) | 60 | 61 | 47
Participants
  Freedom from recurrent VT | 41 | 30 | 32
  Experienced recurrent VT | 19 | 31 | 15

3. Secondary Outcome: Freedom From Cardiovascular Rehospitalization
Description: Cardiovascular rehospitalization is defined as a hospital admission after the randomized procedure for heart failure, procedure-associated complication, or arrhythmia-related causes during the follow-up period.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | ICD With Ablation | ICD Only | Ablation Only (Registry)
Number analyzed (Participants) | 60 | 61 | 47
Participants
  Freedom from cardiovascular rehospitalization | 43 | 41 | 35
  Experienced cardiovascular rehospitalization | 17 | 20 | 12

4. Secondary Outcome: Freedom From All-cause Mortality
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | ICD With Ablation | ICD Only | Ablation Only (Registry)
Number analyzed (Participants) | 60 | 61 | 47
Participants
  Freedom from all-cause mortality | 55 | 57 | 44
  Experienced all-cause mortality | 5 | 4 | 3

5. Other Pre Specified Outcome: Comparison of Outcomes in Ablation Only Registry With Randomized Patients
Time Frame: 2 years
Measure: Number; unit: participants
Groups:
- Randomized Groups (ICD With Ablation and ICD Only): Subjects who meet inclusion/exclusion criteria will be entered into the randomized trial. Randomization will be 1:1 between control group and ablation group. Those randomized to the control group will receive ICD therapy and routine drug therapy (including antiarrhythmic drugs as indicated). Subjects randomized to the ablation group will receive ablation therapy plus ICD for ventricular tachycardia.
- Registry (Ablation Only): The registry will enroll patients who refuse an implantable cardioverter defibrillator (ICD) and are thus not randomized. This arm will assess the efficacy of catheter ablation in the absence of background ICD therapy.
  Catheter Ablation: Catheter ablation is a procedure that uses radiofrequency energy to destroy a small area of heart tissue that is causing rapid and irregular heartbeats. Destroying this tissue helps restore the heart's regular rhythm.
Arm/Group | Randomized Groups (ICD With Ablation and ICD Only) | Registry (Ablation Only)
Number analyzed (Participants) | 121 | 47
participants
  Recurrence of VT | 50 | 15
  Cardiovascular Rehospitalization | 37 | 12
  All-Cause Mortality | 9 | 3

ADVERSE EVENTS:
Time Frame: Subjects were followed for a mean of 2 years, and up to a maximum of 5 years.
Arm/Group | ICD With Ablation | ICD Only | Ablation Only (Registry)
All-Cause Mortality (participants affected / at risk) | 5/60 | 4/61 | 3/47
Serious Adverse Events (participants affected / at risk) | 20/60 | 20/61 | 15/47
Other Adverse Events (participants affected / at risk) | 19/60 | 31/61 | 15/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ICD With Ablation (N=60) | ICD Only (N=61) | Ablation Only (Registry) (N=47)
Procedure Complication (Cardiac disorders) | 5 | 0 | 1
Rehospitalization (Cardiac disorders) | 17 | 20 | 12
Mortality (Cardiac disorders) | 5 | 4 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ICD With Ablation (N=60) | ICD Only (N=61) | Ablation Only (Registry) (N=47)
Arrhythmia, Palpitation (Cardiac disorders) | 19 | 31 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT02848781/Prot_SAP_000.pdf
  • Informed Consent Form (2016-01-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT02848781/ICF_001.pdf